CLINICAL TRIAL: NCT04419168
Title: Cognitive Behavioral Therapy and Real-Time Pain Management Intervention for Sickle Cell Via Mobile Applications
Acronym: CaRISMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kaleab Abebe, PhD, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20110346; CER-2018C2-13320 20 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2020-05-28; First posted 2020-06-05 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pain; Depression, Anxiety; Opioid Use
Keywords: sickle cell disease; pain; opioids; depression; cognitive behavioral therapy; mobile technology; digital health; mHealth; implementation science; community-based participatory research
MeSH Terms: conditions — Chronic Pain; Depression; Anxiety Disorders; Anemia, Sickle Cell; Pain

STUDY DESIGN:
Intervention Model Description: comparative effectiveness trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cCBT (Experimental): Computerized cognitive behavioral therapy (cCBT) for pain. The cCBT program will teach users how to recognize negative thoughts and emotions, use cognitive skills and problem-solving, and apply coping behaviors such as distraction, activity scheduling, and relaxation. The cCBT arm emphasizes skills acquisition and learning through practice; this intervention is consistent with the tailored behavioral services patients would receive individually or as a group when working with a psychologist or behavioral pain specialist.
  Interventions: Other: cCBT
- m-Education (Experimental): Mobile-delivered pain and sickle cell disease education (m-Education). The m-Education program will teach users about chronic pain, healthy lifestyle tips (e.g., nutrition and exercise), and facts about SCD. This program is consistent with the education patients and families would receive with a patient educator.
  Interventions: Other: m-Education

INTERVENTIONS:
Other: cCBT — A digital, internet-delivered, evidence-based chatbot programmed to deliver content for both cCBT.
  Arms: cCBT
Other: m-Education — A digital, internet-delivered, evidence-based chatbot programmed to deliver content for both m-Education.
  Arms: m-Education

SUMMARY:
The investigators are conducting a comparative effectiveness trial among adult patients with sickle cell disease (SCD) who report chronic pain (N = 350), randomized to receive either mobile phone-delivered computerized cognitive behavioral therapy (cCBT; n = 175) or digital education (m-Education; n = 175). Both intervention groups will receive weekly (more frequent if requested or needed) follow-up with a health coach for at least 3 months to reinforce learned materials. Both groups will also use their mobile device to track daily pain, mood, and medication used for two-week periods at baseline and each of the follow-up points (3, 6 and 12 months). Participants will also be given access to a study-associated online support group page where members can discuss with other patients, issues participants faced and what skills were or could be used to address them. Participants will continue all routine care including opioid pain management and novel therapies.

DETAILED DESCRIPTION:
CaRISMA is a randomized comparative effectiveness trial among adult patients with SCD who report chronic pain (N = 350) randomized to receive either cCBT (n = 175) or m-Education (n = 175). A third group of adult patients with SCD who do not meet the criteria for having chronic pain or who are not interested in participating in the intervention will be a convenience non-chronic pain comparison group and will not receive any intervention or scheduled follow-up. The non-chronic pain comparison group will only complete the battery of questionnaires at baseline and each time they return to the clinic for a medical visit. The study will access patients' stored information or verbally obtained information to assess a person's eligibility and suitability for potential participation in the study.

All adult patients, age 18 or above, with a self-report SCD diagnosis, are willing to complete a brief stress and pain functioning screener (stress/pain screener). The stress/pain screener includes measures of depression, anxiety, disability, pain (intensity, quality, and location), and quality of life. The PHQ-9 and GAD-7 measures are administered as part of routine clinical care at the UPMC comprehensive sickle cell clinic and will both be utilized as part of the stress and pain functioning screener for research purposes in the study. Each patient completes electronic versions of all or some of these scales before the sickle cell clinic social worker or psychologist sees them. The total screener typically takes patients about 15-20 minutes to complete.

Patients who do meet the criteria for having chronic pain will be randomized to one of the two intervention groups. For at least 12 weeks, one group will be asked to engage in a mobile cCBT program tailored for adults with SCD. The second group will receive pain and SCD education on mobile phones (m-Education). Both programs use identical mobile technology platforms; only the content differs. The cCBT program focuses on teaching behavioral coping skills through participants' "seeing and doing" while the pain education arm focuses on improving self-management through participants' "learning and knowing" more about pain and SCD. All participants in the intervention group will have weekly follow-ups with a health coach and will track pain symptoms daily during the intervention. A smartphone is required to participate in the intervention. If an interested and eligible participant does not have a smartphone, one may be provided to them. Upon completion of the study, the participant may keep the phone after completing all study elements, including having the study team remove all study-related data from the phone.

Both arms of the intervention will be delivered through pre-programmed chatbot interactions administered in a mobile messaging app. The intervention arm is automatically assigned via the chatbot. When the CaRISMA intervention is opened for the first time, it will automatically randomize each participant to either study arm: cCBT or m-Education. The participants will not know which arm they have been assigned to, and they will only have access to the materials included in the respective study arm

Participants will receive a link to our online survey tool where they will be asked to respond to a set of questionnaires and Painimation, a novel pain assessment tool.

The questionnaires are as follows: Sickle Cell Self-Efficacy Scale (SCSS), Patient- Reported Outcomes Measurement Information System (PROMIS) Pain Interference, Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-ME), Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorders Scale (GAD- 7), and the Current Opioid Misuse Measure (COMM). For participants who are eligible to be randomized, in addition to baseline questionnaires, items from the Coping Strategies Questionnaire (CSQ) will be asked through the messaging app as participants progress through their respective programs.

The Painimation tool is an electronic pain assessment tool developed by our team at the University of Pittsburgh that allows users to better communicate their pain symptoms. Patients are provided with a selection of animations that they use to describe the quality of their pain. The animations can be increased or decreased in speed, color saturation, focus, and size, to reflect the intensity of their pain.

For intervention participants, in addition to the quantitative assessments, our partners at the Qualitative, Evaluation, And Stakeholder Engagement (Qual EASE) Research Services will conduct a set of qualitative interviews to further understand which intervention works best for whom and when, the lived experience of patients in the trial, and differences in perceptions between depression subgroups. Qual- EASE will randomly select 48 participants (of the 350) to be interviewed. Attending the qualitative interviews is completely voluntary and participants may opt out at any time. However, if one of the 48 selected participants does opt out, Qual-EASE will invite another participant, of those not previously selected, as a replacement.

In the first three months of the study, intervention participants will complete all modules of their assigned study arm (cCBT or m-Education) at their own pace. The recommended progression is one module per week; this will give participants time to practice the techniques taught in each module. Participants will be asked to complete a daily electronic diary to track their pain symptoms. Only intervention arm participants will receive follow-up assessment. The convenience comparison group will not be followed with scheduled assessments.

At the 3-month assessment (T1) (i.e., three months after enrollment, on the same date the participant began the study) participants will again receive a link to our online survey tool to complete the second iteration of Painimation, the SCSS, PROMIS, ASCQ-ME, PHQ-9 and GAD-7. If participants have questions while completing these questionnaires, they may contact their health coach for guidance.

Participants will also be asked to complete daily pain intensity entries in the electronic diary. If participants do not complete the questionnaires or the pain intensity entries, health coaches will contact them and remind them to do so. The 48 patients selected for qualitative interviews will have their second interview with Qual- EASE at this time.

Between months 4-6, participants will continue to use the CaRISMA intervention but will no longer have weekly follow-ups with a health coach except upon request or on an as-needed basis. At the end of month 6 (T2), they will receive a link to our online survey tool to complete Painimation, the SCSS, PROMIS, ASCQ-ME, PHQ-9, and GAD-7 for the third time. Participants will continue to complete daily pain intensity entries through the electronic diary.

Between months 6-12, participants will continue daily pain diary submissions and communication with health coaches only as desired. Additionally, Qual-EASE will conduct the final set of qualitative interviews with 48 of the 350 participants.

In the final month of the study (T3), participants will receive a link to our online survey tool to complete Painimation, the SCSS, PROMIS, ASCQ-ME, PHQ-9, GAD- 7 and COMM for the final time.

The pain diary may include some version of the following types of questions in daily assessments:

* Using any number from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable, what is your pain level today?
* Did you take opiate medications today?
* Which one of the following emojis best represents your mood today? The pain diary may include some version of the following types of questions in weekly assessments:
* Using any number from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable, what is your pain level today?
* Did you take opiate medications today?
* Compared to what you used yesterday, is the amount of opiate meds you took today less than yesterday, the same as yesterday, or more than yesterday?
* Did you take non-opiate medications today?
* This past week, how often have you been bothered by little interest or pleasure in doing things?
* This past week, how often have you been bothered by feeling down, depressed, or irritable?
* This past week, how often have you been bothered by feeling nervous, anxious, or on edge?
* This past week, how often have you been bothered by not being able to stop or control worry?

Medical Outcomes (PCORnet). For patients recruited at one of the five clinical sites, we will evaluate objectively measured opioid medication refills and emergency department visits or hospitalizations for pain crisis. We will be working in collaboration with PCORnet to collect data retrospectively (from the past 12 months) and prospectively (12 months from the date of enrollment) from patient medical records.

These data will allow us to track medications including opioid pain medication prescriptions and refills, and health care utilization (i.e., emergency department visits and hospitalizations), as well as lab values (e.g., hemoglobin level) and clinical outcomes (e.g., end-organ damage score). For the patients recruited from our community partner organizations or online who are not affiliated with a participating clinical center, we will only acquire or evaluate their medical records for the purpose of confirming their sickle cell diagnosis.

The primary outcome is the change in pain interference at 6 months. Secondary outcomes include changes in pain intensity, depression (PHQ), anxiety (GAD), quality of life (ASCQ-ME), self-efficacy (SCSES), opioid misuse (COMM), and health care utilization at 6 and 12 months. The study team has updated the outcomes to be more comprehensive due to the funder's requirement that it align with the contract milestones

ELIGIBILITY:
Inclusion Criteria:

* People with any type of sickle cell disease
* Male or female, age 18 years or older
* Reports chronic pain: i.e pain more days that not for the past 3 months or longer and/or is prescribed daily or long-acting opioids for pain.
* English speaking

Exclusion Criteria:

* Any potential participants who fail consent comprehension questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Illinous-Chicago, Chicago, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oluwole OB, McGill LS, Gayle K, O'Brien JA, Abebe KZ, Jonassaint CR, Hamm M. Experiences With a Multicomponent Digital Behavioral Pain Management Intervention for Adults With Sickle Cell Disease: Qualitative Analysis of the CaRISMA Trial. JMIR Hum Factors. 2025 Aug 5;12:e73719. doi: 10.2196/73719. PMID 40763347
- [Derived] Jonassaint CR, Parchuri E, O'Brien JA, Lalama CM, Lin J, Badawy SM, Hamm ME, Stinson J, Lalloo C, Carroll CP, Saraf SL, Gordeuk VR, Cronin R, Shah N, Lanzkron SM, Liles D, Trimnell C, Bailey L, Lawrence RH, Abebe KZ. Mental health, pain and likelihood of opioid misuse among adults with sickle cell disease. Br J Haematol. 2024 Mar;204(3):1029-1038. doi: 10.1111/bjh.19243. Epub 2024 Jan 3. PMID 38171495
- [Derived] Badawy SM, Abebe KZ, Reichman CA, Checo G, Hamm ME, Stinson J, Lalloo C, Carroll P, Saraf SL, Gordeuk VR, Desai P, Shah N, Liles D, Trimnell C, Jonassaint CR. Comparing the Effectiveness of Education Versus Digital Cognitive Behavioral Therapy for Adults With Sickle Cell Disease: Protocol for the Cognitive Behavioral Therapy and Real-time Pain Management Intervention for Sickle Cell via Mobile Applications (CaRISMA) Study. JMIR Res Protoc. 2021 May 14;10(5):e29014. doi: 10.2196/29014. PMID 33988517

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | cCBT | m-Education
Started | 181 | 178
3-month Follow up Visit | 134 | 135
Completed | 125 | 125
Not Completed | 56 | 53
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 7 | 7
Not completed — Missed 6-month Visit | 48 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | cCBT | m-Education | Total
Number analyzed (Participants) | 181 | 178 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (9.9) | 36.3 (11.1) | 36.3 (10.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Biological Sex: Male | 69 | 49 | 118
  Biological Sex: Female | 111 | 128 | 239
  Biological Sex: Prefer not to answer | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 15
  Not Hispanic or Latino | 156 | 152 | 308
  Unknown or Not Reported | 19 | 17 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 169 | 163 | 332
  White | 0 | 2 | 2
  More than one race | 7 | 8 | 15
  Unknown or Not Reported | 5 | 4 | 9
PROMIS Pain Interference [Mean (Standard Deviation); unit: T-score] — The 8-item Patient Reported Outcomes Measure Information System Pain Interference (PROMIS-8a) assesses the effect of patient-reported pain on relevant aspects of a person's life and may include the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities in the past 7 days. The items use 1-5 Likert scale with higher scores indicating greater pain interference. The raw total score (ranging from 8 to 40) is transformed using a T-score for a mean of 50, standard deviation of 10, in referent population. Higher T-scores indicate greater pain.
  T-score | 62.2 (7.3) | 62.9 (7) | 62.6 (7.1)
Average pain intensity [Mean (Standard Deviation); unit: units on a scale] — At each timepoint, participants will be asked to enter their daily pain via a mobile website for 2 weeks. The mean pain intensity is calculated during this 2 week period and used for analyses. Pain ratings range from 0-10 where 0 is no pain and 10 is the worst pain imaginable. Population: Only participants who completed the pain diary were included.
  units on a scale
    number analyzed (Participants) | 151 | 148 | 299
    (all) | 4.2 (2.5) | 4.5 (2.5) | 4.4 (2.5)
Patient Health Questionnaire (PHQ) [Mean (Standard Deviation); unit: units on a scale] — PHQ-9 assesses the degree of depression severity. The PHQ-9 total score is for nine items, all rated as 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 27. Scores of 5, 10, 15, and 20 represent cut-off points for mild, moderate, moderately severe, and severe depression, respectively Population: Only participants who scored >0 on PHQ-2 (first two items of the PHQ) were administered the rest of the survey.
  units on a scale
    number analyzed (Participants) | 144 | 148 | 292
    (all) | 11 (5) | 10 (5) | 10 (5)
Generalized Anxiety Disorder Scale [Mean (Standard Deviation); unit: units on a scale] — GAD-7 evaluates the severity of anxiety. The GAD-7 total score for the 7 items ranges from 0 to 21. Scores of 5, 10, and 15 represent the cut-off points for mild, moderate, and severe anxiety, respectively. Population: Only participants who scored >0 on GAD-2 (first two items of the GAD) were administered the rest of the survey.
  units on a scale
    number analyzed (Participants) | 131 | 120 | 251
    (all) | 9 (5) | 9 (5) | 9 (5)
Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-ME) [Mean (Standard Deviation); unit: T-score] — The ASCQ-ME emotional functioning and social impact quality-of-life measure was specifically designed for SCD and evaluates the health care experience of patients with SCD, emotional response to stress, and social relationships. For each subscale (emotional impact and social functioning impact), there are 5 questions using a 1-5 Likert scale with lower scores indicating worse health. Raw total scores (ranging from 5 to 25) are transformed using a T-score for a mean of 50, standard deviation of 10, in referent population. Lower T-scores indicate worse health.
  T-score
    Social Functioning | 47.4 (8.6) | 47.1 (7.1) | 47.3 (7.9)
    Emotional Impact | 47.2 (8.8) | 48.8 (8.8) | 48.0 (8.8)
Sickle Cell Self-Efficacy Scale (SCSES) [Mean (Standard Deviation); unit: units on a scale] — The Sickle Cell Disease Self-Efficacy Scale is a nine-item self-administered questionnaire that measures disease-specific perceptions of the ability to manage day-to-day issues resulting from sickle cell disease (SCD). Items are scores according to a five-point scale ranging from "1 - Not sure at all" to "5 - Very sure." Responses from individual items are summed to give an overall score with higher scores indicating greater self-efficacy (ranging from 9 to 45).
  units on a scale | 28 (6) | 29 (7) | 29 (7)
Total Body Area Shaded (Painimation) [Mean (Standard Deviation); unit: mean percentage of total body area shade] — Painimation is an electronic pain assessment tool that allows users to better communicate pain symptoms. Patients are provided with a selection of animations (painimations) that they use to describe the quality of their pain. For each participant, there are 22 body sections that can be shaded to show where they have pain. To get the percent of total body area shaded across all sections of the body, the sum of the body area shaded for each section of the body (numerator) was divided by the sum of the total body area of each section that could be shaded (denominator).
  mean percentage of total body area shade | 13 (14.7) | 14 (15.4) | 13.5 (15.0)
Current Opioid Misuse Measure (COMM) [Mean (Standard Deviation); unit: units on a scale] — Current Opioid Misuse Measure (COMM) is a self-report measure to monitor indicators of current aberrant drug-related behaviors in patients with chronic pain on opioid therapy. Total scores are summed across the 9 individual items and range from 0-36, with higher scores representing greater misuse.
  units on a scale | 9 (6) | 8 (5) | 9 (5)

OUTCOME MEASURES:

1. Primary Outcome: 6-month Change in PROMIS Pain Interference
Description: The 8-item Patient Reported Outcomes Measure Information System Pain Interference (PROMIS-8a) assesses the effect of patient-reported pain on relevant aspects of a person's life and may include the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities in the past 7 days. The items use 1-5 Likert scale with higher scores indicating greater pain interference. The raw total score (ranging from 8 to 40) is transformed using a T-score for a mean of 50, standard deviation of 10, in referent population. Higher T-scores indicate greater pain.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 181 | 178
T-score | -2.13 [-3.42 to -0.84] | -2.66 [-3.97 to -1.36]
Statistical Analysis 1: Comparison: cCBT vs m-Education; Test type: Superiority; p = .57, Mixed Models Analysis; Mean Difference (Final Values) = .54, 95% CI 2-sided [-1.30 to 2.37]

2. Secondary Outcome: 6-month Change in Daily Pain Intensity
Description: At each timepoint, participants will be asked to enter their daily pain via a mobile website for 2 weeks. The mean pain intensity is calculated during this 2 week period and used for analyses. Pain ratings range from 0-10 where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: Baseline and 6 months
Population: Analysis population consisted of randomization participants with sufficient pain diary data over the 2 week period after each visit.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 151 | 148
score on a scale | 0.20 [-0.18 to 0.58] | 0.13 [-0.25 to 0.51]
Statistical Analysis 1: Comparison: cCBT vs m-Education; Test type: Superiority; p = 0.79, Mixed Models Analysis; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.46 to 0.61]

3. Secondary Outcome: 6-month Change in Patient Health Questionnaire (PHQ)
Description: PHQ-9 assesses the degree of depression severity. The PHQ-9 total score is for nine items, all rated as 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 27. Scores of 5, 10, 15, and 20 represent cut-off points for mild, moderate, moderately severe, and severe depression, respectively.
Time Frame: Baseline and 6 months
Population: Analysis population consisted of randomization participants with PHQ2>0.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 144 | 148
score on a scale | -1.33 [-2.28 to -0.39] | -1.12 [-2.06 to -0.18]
Statistical Analysis 1: Comparison: cCBT vs m-Education; Test type: Superiority; p = 0.75, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-1.55 to 1.12]

4. Secondary Outcome: 6-month Change in Generalized Anxiety Disorder Scale-7 (GAD-7)
Description: GAD-7 evaluates the severity of anxiety. The GAD-7 total score for the 7 items ranges from 0 to 21. Scores of 5, 10, and 15 represent the cut-off points for mild, moderate, and severe anxiety, respectively.
Time Frame: Baseline and 6 months
Population: Analysis population consisted of randomization participants with GAD2>0.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 131 | 120
score on a scale | -0.85 [-1.68 to -0.01] | -1.49 [-2.40 to -0.58]
Statistical Analysis 1: Comparison: cCBT vs m-Education; Test type: Superiority; p = 0.31, Mixed Models Analysis; Mean Difference (Final Values) = 0.64, 95% CI 2-sided [-0.60 to 1.87]

5. Secondary Outcome: 6-month Change in Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-ME)
Description: The ASCQ-ME emotional functioning and social impact quality-of-life measure was specifically designed for SCD and evaluates the health care experience of patients with SCD, emotional response to stress, and social relationships. For each subscale (emotional impact in the past 7 days and social functioning impact in the past 30 days), there are 5 questions using a 1-5 Likert scale with lower scores indicating worse health. Raw total scores (ranging from 5 to 25) are transformed using a T-score for a mean of 50, standard deviation of 10, in referent population. Lower T-scores indicate worse health.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 181 | 178
T-score
  ASCQ-ME Social Functioning Impact | 2.45 [1.13 to 3.76] | 2.34 [1.00 to 3.68]
  ASCQ-Me Emotional Impact | 3.51 [2.29 to 4.73] | 1.79 [0.55 to 3.04]
Statistical Analysis 1: Comparison: cCBT vs m-Education; These results correspond to ASCQ-Me Social Functioning Impact only; Test type: Superiority; p = 0.91, Mixed Models Analysis; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-1.77 to 1.99]
Statistical Analysis 2: Comparison: cCBT vs m-Education; These results correspond to ASCQ-Me Emotional Impact only; Test type: Superiority; p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 1.72, 95% CI 2-sided [-0.03 to 3.46]

6. Secondary Outcome: 6-month Change in Sickle Cell Self-Efficacy Scale (SCSES)
Description: The Sickle Cell Disease Self-Efficacy Scale is a nine-item self-administered questionnaire that measures disease-specific perceptions of the ability to manage day-to-day issues resulting from sickle cell disease (SCD). Items are scores according to a five-point scale ranging from "1 - Not sure at all" to "5 - Very sure." Responses from individual items are summed to give an overall score with higher scores indicating greater self-efficacy (ranging from 9 to 45).
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 181 | 178
score on a scale | 1.45 [0.44 to 2.46] | 0.32 [-0.70 to 1.35]
Statistical Analysis 1: Comparison: cCBT vs m-Education; Test type: Superiority; p = 0.12, Mixed Models Analysis; Mean Difference (Final Values) = 1.13, 95% CI 2-sided [-0.31 to 2.56]

7. Secondary Outcome: Change From Baseline in Percent of Total Body Area Shaded (Painimation) at 6 Months
Description: Painimation is an electronic pain assessment tool that allows users to better communicate pain symptoms. Patients are provided with a selection of animations (painimations) that they use to describe the quality of their pain. The painimations can be adjusted to reflect pain intensity. Screenshots of the Painimation app illustrate the splash screen, paintable body image, and selection of painimations to indicate the quality and intensity of pain. A higher mean % is indicative of greater pain. For analyses, mean percentages are transformed via arc-sine square in order to normalize.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: percentage of total body area shaded
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 181 | 178
percentage of total body area shaded | -0.0338 [-0.0633 to -0.0042] | -0.0314 [-0.0611 to -0.0016]
Statistical Analysis 1: Comparison: cCBT vs m-Education; Test type: Superiority; p = 0.91, Mixed Models Analysis; Mean Difference (Final Values) = -0.0024, 95% CI 2-sided [-0.0443 to 0.0395]

8. Secondary Outcome: 12-month Change in PROMIS Pain Interference
Description: as for outcome 1
Time Frame: Baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 181 | 178
T-score | -1.50 [-2.94 to -0.07] | -1.93 [-3.39 to -0.47]
Statistical Analysis 1: Comparison: cCBT vs m-Education; Test type: Superiority; p = 0.68, Mixed Models Analysis; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-1.61 to 2.48]

9. Secondary Outcome: 12-month Change in Daily Pain Intensity
Description: as for outcome 2
Time Frame: Baseline and 12 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 151 | 148
score on a scale | 0.06 [-0.31 to 0.44] | -0.02 [-0.42 to 0.37]
Statistical Analysis 1: Comparison: cCBT vs m-Education; Test type: Superiority; p = 0.75, Mixed Models Analysis; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.46 to 0.63]

10. Secondary Outcome: 12-month Change in Patient Health Questionnaire (PHQ)
Description: as for outcome 3
Time Frame: Baseline and 12 months
Population: PHQ-9 for Clinic participants and PHQ-8 for Virtual participants with baseline PHQ-2 >0
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 144 | 148
score on a scale | -1.34 [-2.39 to -0.29] | -0.24 [-1.24 to 0.77]
Statistical Analysis 1: Comparison: cCBT vs m-Education; Test type: Superiority; p = 0.14, Mixed Models Analysis; Mean Difference (Final Values) = -1.10, 95% CI 2-sided [-2.56 to 0.35]

11. Secondary Outcome: 12-month Change in Generalized Anxiety Disorder Scale-7 (GAD-7)
Description: as for outcome 4
Time Frame: Baseline and 12 months
Population: GAD-7 for all participants with baseline GAD-2 >0
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 131 | 120
score on a scale | -0.70 [-1.69 to 0.29] | -0.46 [-1.52 to 0.59]
Statistical Analysis 1: Comparison: cCBT vs m-Education; Test type: Superiority; p = 0.75, Mixed Models Analysis; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-1.69 to 1.21]

12. Secondary Outcome: 12-month Change in Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-ME)
Description: as for outcome 5
Time Frame: Baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 181 | 178
T-score
  ASCQ-Me Social Functioning Impact | 2.31 [0.91 to 3.72] | 1.61 [0.17 to 3.04]
  ASCQ-Me Emotional Impact | 3.03 [1.71 to 4.34] | 1.03 [-0.31 to 2.37]
Statistical Analysis 1: Comparison: cCBT vs m-Education; These results correspond to ASCQ-Me Social Functioning Impact only; Test type: Superiority; p = 0.49, Mixed Models Analysis; Mean Difference (Final Values) = 0.71, 95% CI 2-sided [-1.30 to 2.71]
Statistical Analysis 2: Comparison: cCBT vs m-Education; These results correspond to ASCQ-Me Emotional Impact only; Test type: Superiority; p = 0.037, Mixed Models Analysis; Mean Difference (Final Values) = 2.00, 95% CI 2-sided [0.12 to 3.88]

13. Secondary Outcome: 12-month Change in Sickle Cell Self-Efficacy Scale (SCSES)
Description: as for outcome 6
Time Frame: Baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 181 | 178
score on a scale | 1.50 [0.40 to 2.61] | -0.63 [-1.75 to 0.50]
Statistical Analysis 1: Comparison: cCBT vs m-Education; Test type: Superiority; p = 0.008, Mixed Models Analysis; Mean Difference (Final Values) = 2.13, 95% CI 2-sided [0.56 to 3.71]

14. Secondary Outcome: 12-month Change in Current Opioid Misuse Measure (COMM)
Description: Current Opioid Misuse Measure (COMM) is a self-reported measure to monitor indicators of current aberrant drug-related behaviors in patients with chronic pain on opioid therapy. Total scores are summed across the 9 individual items and range from 0-36, with higher scores representing greater misuse.
Time Frame: Baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 181 | 178
score on a scale | -1.72 [-2.54 to -0.91] | -1.38 [-2.21 to -0.55]
Statistical Analysis 1: Comparison: cCBT vs m-Education; Test type: Superiority; p = 0.56, Mixed Models Analysis; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-1.51 to 0.82]

15. Secondary Outcome: Change From Baseline in Percent of Total Body Area Shaded (Painimation) at 12 Months
Description: as for outcome 7
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: percentage of total body area shaded
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 181 | 178
percentage of total body area shaded | -0.05 [-0.08 to -0.02] | -0.05 [-0.08 to -0.02]
Statistical Analysis 1: Comparison: cCBT vs m-Education; Test type: Superiority; p = 0.95, Mixed Models Analysis; Mean Difference (Final Values) = -0.0013, 95% CI 2-sided [-0.0464 to 0.0437]

16. Secondary Outcome: Number of Opioid Prescriptions
Description: For patients recruited at one of the six clinical sites, study team will evaluate objectively measured opioid medication prescriptions and refills. Study team will work in collaboration with PCORnet to collect outcome data 12 months after enrollment from patients' electronic health records.
Time Frame: 12 months
Population: Analysis population consisted of randomization participants with available data from PCORnet.
Measure: Number (95% Confidence Interval); unit: Prescriptions per person-year
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 200 | 200
Prescriptions per person-year | 30.15 [23.97 to 37.91] | 27.19 [21.77 to 33.95]
Statistical Analysis 1: Comparison: cCBT vs m-Education; Test type: Superiority; p = 0.49, Negative Binomial Regression; Adjustments were made for clinic site, baseline depression (high vs low), and corresponding health care use in the 12 months prior to study entry; Incidence Rate Ratio = 1.11, 95% CI 2-sided [0.83 to 1.48]

17. Secondary Outcome: Number of Emergency Department Visits
Description: For patients recruited at one of the six clinical sites, study team will evaluate objectively measured emergency department visits. Study team will work in collaboration with PCORnet to collect outcome data 12 months after enrollment from patients' electronic health records.
Time Frame: 12 months
Population: Analysis population consisted of randomization participants with available data from PCORnet.
Measure: Number (95% Confidence Interval); unit: ED visits per person-year
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 200 | 200
ED visits per person-year | 2.65 [1.92 to 3.66] | 1.86 [1.34 to 2.59]
Statistical Analysis 1: Comparison: cCBT vs m-Education; Test type: Superiority; p = 0.10, Negative Binomial Regression; [statistical method as in outcome 16, analysis 1]; Incidence Rate Ratio = 1.43, 95% CI 2-sided [0.93 to 2.18]

18. Secondary Outcome: Number of Hospitalizations
Description: For patients recruited at one of the six clinical sites, study team will evaluate objectively measured hospitalizations. Study team will work in collaboration with PCORnet to collect outcome data 12 months after enrollment from patients' electronic health records.
Time Frame: 12 months
Population: Analysis population consisted of randomization participants with available data from PCORnet.
Measure: Number (95% Confidence Interval); unit: Hospitalizations per person-year
Arm/Group | cCBT | m-Education
Number analyzed (Participants) | 200 | 200
Hospitalizations per person-year | 1.16 [0.83 to 1.62] | 0.89 [0.64 to 1.23]
Statistical Analysis 1: Comparison: cCBT vs m-Education; Test type: Superiority; p = 0.22, Negative Binomial Regression; [statistical method as in outcome 16, analysis 1]; Incidence Rate Ratio = 1.31, 95% CI 2-sided [0.85 to 2.03]

ADVERSE EVENTS:
Time Frame: 1 year.
Arm/Group | cCBT | m-Education
All-Cause Mortality (participants affected / at risk) | 3/181 | 1/178
Serious Adverse Events (participants affected / at risk) | 3/181 | 1/178
Other Adverse Events (participants affected / at risk) | 0/181 | 0/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cCBT (N=181) | m-Education (N=178)
General disorders and administration site conditions (General disorders) | 3 (3) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT04419168/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT04419168/SAP_001.pdf